CLINICAL TRIAL: NCT01053962
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled, 14-Day Repeat, Oral, Dose Ranging Study to Assess the Safety, Pharmacokinetic and Pharmacodynamic Effects of SP-304 in Patients With Chronic Idiopathic Constipation
Brief Title: SP-304 Dose Ranging Study in Patients With Chronic Idiopathic Constipation
Acronym: CIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP-SP304201-09
Record Dates: First submitted 2010-01-12; First posted 2010-01-22 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Chronic Idiopathic Constipation
Keywords: Chronic Idiopathic Constipation; Constipation; Irritable Bowel Syndrome
MeSH Terms: conditions — Constipation; Irritable Bowel Syndrome | interventions — plecanatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- SP-304 0.3 mg (Experimental): SP-304 0.3 mg tablet by mouth once daily for 14 consecutive days.
  Interventions: Drug: SP-304 0.3 mg
- SP-304 1.0 mg (Experimental): SP-304 1.0 mg tablet by mouth once daily for 14 consecutive days.
  Interventions: Drug: SP-304 1.0 mg
- SP-304 3.0 mg (Experimental): SP-304 3.0 mg tablet by mouth once daily for 14 consecutive days
  Interventions: Drug: SP-304 3.0 mg
- SP-304 9.0 mg (Experimental): SP-304 9.0 mg tablet by mouth once daily for 14 consecutive days.
  Interventions: Drug: SP-304 9.0 mg
- Placebo (Placebo Comparator): Placebo tablet by mouth once daily for 14 consecutive days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SP-304 0.3 mg — SP-304 0.3 mg
  Arms: SP-304 0.3 mg
Drug: SP-304 1.0 mg — SP-304 1.0 mg
  Arms: SP-304 1.0 mg
Drug: SP-304 3.0 mg — SP-304 3.0 mg
  Arms: SP-304 3.0 mg
Drug: SP-304 9.0 mg — SP-304 9.0 mg
  Arms: SP-304 9.0 mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a Phase 2a, randomized, double-blind, placebo-controlled, 14-day repeat oral, dose ranging study to determine the safety, pharmacokinetics (PK) and pharmacodynamics (PD) effects of SP-304 in patients with chronic idiopathic constipation.

DETAILED DESCRIPTION:
This is a Phase 2a, randomized, double-blind, placebo-controlled, 14-day repeat oral, dose ranging study to determine the safety, PK and PD effects of SP-304 in patients with chronic idiopathic constipation. Patients diagnosed with chronic idiopathic constipation (CIC) will be screened for the anticipated 4 cohorts, to yield 80 randomized patients for enrollment. Four dose cohorts are planned (0.3 mg, 1.0 mg, 3.0mg, and 9.0 mg) with 20 patients per dose cohort [randomization ratio 3:1 (15 receive SP-304:5 receive placebo)]. Patients who continue to meet all the entry criteria and complete the pre-treatment bowel movement (BM) diary will receive, in a double-blind, randomized fashion, SP-304 or matching placebo. It is expected that each patient will complete all 14 days of dosing (including making accurate BM diary entries for all 14 days in the treatment period). All patients receiving at least one dose of SP-304 or matching placebo will be considered evaluable for the safety endpoints. If a patient receives at least 5 doses per treatment week (1 dose per day for 7 days) and has completed BM diary entries for those 5 dosing days in each corresponding treatment week, he/she will be considered evaluable.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to understand and willing to sign the Informed Consent Form (ICF) and capable of providing written authorization for use and disclosure of protected health information per requirements of 45 CFR 164.508 (Health Insurance Portability and Accountability Act [HIPAA]).
* Subject is male or non-pregnant, non-breastfeeding female, between 18 and 75 years of age (inclusive) at the time of first dose.
* Subject has a body mass index (BMI) between 18 and 35 kg/m2.
* Subject meets the Rome III Diagnostic Criteria for constipation (Drossman, 2006) for the past 3 months with symptom onset > 6 months prior to diagnosis.

Exclusion Criteria:

* Subject reports loose stool (fluffy pieces with ragged edges, a mushy stool) or watery stool (no solid pieces, entirely liquid; BSFS score of 6 or 7, respectively) in the absence of any laxative, enema, suppository or prohibited medicine for > 25% of BMs during the 3 months prior to the Screening visit and during the 14 day pre-treatment period.
* Subjects who meet the Rome III criteria for IBS.
* Subject has failed to complete the pre-treatment bowel movement diary accurately and completely during the pre-treatment period prior to Day 1 dosing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2010-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary S Jacob, Ph.D., Study Director — Synergy Pharmaceuticals Inc.
Locations (14):
- United States (14):
  - Novara Clinical Research, Mesa, Arizona
  - Genova Clinical Research, Tucson, Arizona
  - Advanced Clinical Research, Anaheim, California
  - Advanced Clinical Research, Orange, California
  - A.G.A. Clinical Trials, Hialeah, Florida
  - Miami Ressearch and Associates, Miami, Florida
  - Lee Research Institute, Shawnee Mission, Kansas
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Universtiy of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Memphis Gastroenterology Group, Germantown, Tennessee
  - Nashville Medical Research Institute, Nashville, Tennessee
  - DCOL Center for Clinical Research, Longview, Texas
  - Pioneer Research Solutions, Sugar Land, Texas

REFERENCES:
- [Result] Shailubhai K, Talluto C, Comiskey S, Foss J, Joslyn A, Jacob G. Phase II Clinical Evaluation of SP-304, a Guanylate Cyclase-C Agonist, for Treatment of Chronic Constipation. Am J Gastroenterology 105 (Supp 1): S487, 2010

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted between 3 March 2010 and 26 August 2010 at 14 study centers in the United States. Four dose cohorts were planned (0.3 mg, 1.0 mg, 3.0 mg, and 9.0 mg with 20 patients per dose cohort randomized in a 3:1 ratio [15 pts receive SP-304, 5 pts receive placebo].
Pre-assignment Details: During the pre-treatment period (Study Days -14 though -1), 84 eligible patients completed daily bowel movement diaries to obtain baseline data. Of these, 78 patients (58 and 20 patients for the SP-304 and placebo treatment groups, respectively) received at least one dose of study drug.
Groups:
- SP-304 0.3 mg: Subjects receiving SP-304 0.3 mg for 14 consecutive days.
- SP-304 1.0 mg: Subjects receiving SP-304 1.0 mg for 14 consecutive days
- SP-304 3.0 mg: Subjects receiving SP-304 3.0 mg for 14 consecutive days
- SP-304 9.0 mg: Subjects receiving SP-304 9.0 mg for 14 consecutive days
- Placebo: Subjects receiving Placebo for 14 consecutive days
Period: Pretreatment Period
Arm/Group | SP-304 0.3 mg | SP-304 1.0 mg | SP-304 3.0 mg | SP-304 9.0 mg | Placebo
Started | 14 | 15 | 16 | 17 | 22
Completed | 14 | 14 | 15 | 15 | 20
Not Completed | 0 | 1 | 1 | 2 | 2
Not completed — Withdrew Consent (Patient/PI) | 0 | 0 | 0 | 1 | 2
Not completed — Venipuncture Failure | 0 | 0 | 1 | 0 | 0
Not completed — Failed Urine drug screen Day 1 | 0 | 1 | 0 | 0 | 0
Not completed — Abnormal Lab values Exl 16 | 0 | 0 | 0 | 1 | 0
Period: Treatment Period
Arm/Group | SP-304 0.3 mg | SP-304 1.0 mg | SP-304 3.0 mg | SP-304 9.0 mg | Placebo
Started | 14 | 14 | 15 | 15 | 20
Completed | 13 | 14 | 15 | 15 | 17
Not Completed | 1 | 0 | 0 | 0 | 3
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1
Not completed — Noncompliance with protocol | 1 | 0 | 0 | 0 | 0
Period: Follow-up Period
Arm/Group | SP-304 0.3 mg | SP-304 1.0 mg | SP-304 3.0 mg | SP-304 9.0 mg | Placebo
Started | 13 | 14 | 15 | 15 | 17
Completed | 13 | 14 | 15 | 15 | 17
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: patients who received at least one dose of study medication (population for primary endpoint).
Groups:
- Total: Total of all reporting groups
Arm/Group | SP-304 1.0 mg | SP-304 3.0 mg | SP-304 9.0 mg | Placebo | SP-304 0.3 mg | Total
Number analyzed (Participants) | 14 | 15 | 15 | 20 | 14 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 14 | 17 | 11 | 65
  >=65 years | 2 | 4 | 1 | 3 | 3 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (10.6) | 48.5 (16.17) | 47.3 (12.71) | 47.7 (14.64) | 51.1 (11.95) | 48.9 (13.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 12 | 18 | 12 | 69
  Male | 0 | 2 | 3 | 2 | 2 | 9
Region of Enrollment [Number; unit: participants]
  United States | 14 | 15 | 15 | 20 | 14 | 78
Complete Spontaneous Bowel Movement Frequency [Mean (Standard Deviation); unit: CSBMs per week] — On daily basis during the 14-day pre-treatment period, patients recorded the number of spontaneous bowel movements having the sensation of complete evacuation (Complete Spontaneous Bowel Movement - CSBM). The Baseline Weekly Frequency of CSBMs during the pre-treatment period was calculated total number of CSBMs divided by 2 (the number of weeks in the pre-treatment period).
  CSBMs per week | 0.6 (0.74) | 0.5 (0.92) | 0.4 (0.54) | 0.3 (0.53) | 0.4 (0.53) | 0.4 (0.66)
Spontaneous Bowel Movement Frequency [Mean (Standard Deviation); unit: events per week] — On daily basis during the 14-day pre-treatment period, patients recorded the number of spontaneous bowel movements (SBM). The Baseline Weekly Frequency of SBMs during the pre-treatment period was calculated total number of SBMs divided by 2 (the number of weeks in the pre-treatment period).
  events per week | 2.2 (0.99) | 2.1 (0.93) | 1.9 (0.75) | 2.0 (1.01) | 2.2 (1.12) | 2.1 (0.95)
Stool Consistency (Bristol Stool Form Scale) [Mean (Standard Deviation); unit: units on a scale] — Using a Daily Diary, patients recorded Stool Consistency using the 7-point Bristol Stool Form Scale (BSFS) (1 = separate hard lumps, like nuts; 2 sausage shaped but lumpy; 3 = like a sausage but with cracks on surface; 4 = like a sausage or snake, smooth and soft; 5 = soft blobs with clear-cut edges; 6 = fluffy pieces with ragged edges, a mushy stool; 7 = watery, no solid pieces, entirely liquid).
  units on a scale | 2.6 (0.84) | 1.8 (0.69) | 2.7 (1.56) | 2.6 (1.28) | 2.5 (0.81) | 2.4 (1.13)
Ease of Passage (Straining) [Mean (Standard Deviation); unit: units on a scale] — Using a Daily Diary, patients recorded Ease of Passage (Straining) using the 7-point Ease-of-Passage Scale (1 = manual disimpaction/enema needed, 2 = severe straining, 3 = moderate straining, 4 = mild straining, 5 = no straining, 6 = urgency, 7 = incontinent).
  units on a scale | 2.8 (0.79) | 2.7 (0.61) | 3.0 (0.89) | 3.0 (0.67) | 3.1 (0.64) | 2.9 (0.72)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Incidences of adverse events from Baseline through the end of the Follow-up period.
Time Frame: 21 days: Baseline through Follow-up (Treatment Days 14, 7 days post treatment)
Population: Safety Population: all patients who received at least one dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | SP-304 0.3 mg | SP-304 1.0 mg | SP-304 3.0 mg | SP-304 9.0 mg | Placebo
Number analyzed (Participants) | 14 | 14 | 15 | 15 | 20
Participants | 3 | 6 | 2 | 6 | 4

2. Secondary Outcome: Change From Baseline Overall in Number of Complete Spontaneous Bowel Movements (CSBM)
Description: Using a Daily Diary, patients recorded the number of spontaneous bowel movements having the sensation of complete evacuation (Complete Spontaneous Bowel Movement - CSBM). The total number of spontaneous bowel movements associated with a feeling of complete evacuation were summed and divided by 2 (the number of weeks in treatment). Change was calculated as the difference between the number of the CSBMs at the completion of the 2-week treatment period, versus the 14-day pretreatment baseline.
Time Frame: Study days 1 through 14
Population: Modified-Intent-to-Treat population: All patients who received at least one dose of study medication and had at least one post-baseline diary assessment. One participant in the SP-304 0.3 mg group did not have information about complete evacuation post-baseline.
Measure: Mean (Standard Deviation); unit: CSBMs per week
Groups:
- SP-304 0.3 mg: Subjects receiving SP-304 0.3 mg for 14 consecutive days.
  SP-304 0.3 mg: Subjects receiving SP-304 0.3 mg for 14 consecutive
- SP-304 1.0 mg: Subjects receiving SP-304 1.0 mg for 14 consecutive days
  SP-304: Subjects receiving SP-304 1.0 mg for 14 consecutive days
- SP-304 3.0 mg: Subjects receiving SP-304 3.0 mg for 14 consecutive days
  SP-304: Subjects receiving SP-304 3.0 mg for 14 consecutive days
- SP-304 9.0 mg: Subjects receiving SP-304 9.0 mg for 14 consecutive days
  SP-304: Subjects receiving SP-304 9.0 mg for 14 consecutive days
- Placebo: Subjects receiving Placebo for 14 consecutive days
  Placebo: Subjects receiving Placebo for 14 consecutive days
Arm/Group | SP-304 0.3 mg | SP-304 1.0 mg | SP-304 3.0 mg | SP-304 9.0 mg | Placebo
Number analyzed (Participants) | 13 | 14 | 15 | 15 | 20
CSBMs per week | 1.7 (2.30) | 3.3 (2.85) | 1.8 (3.75) | 2.7 (2.89) | 2.0 (3.02)

3. Secondary Outcome: Change From Baseline Overall in Number of Spontaneous Bowel Movements (SBM)
Description: Using a Daily Diary, patients recorded the number of spontaneous bowel movements (SBM). The overall weekly frequency was calculated as the total number of SBMs divided by 2 (the number weeks of treatment). Change was calculated as the difference between the number of the SBMs at the completion of the 2-week treatment period, versus the 14-day pretreatment baseline.
Time Frame: Study Days 1 through 14
Population: Modified-Intent-to-Treat population: All patients who received at least one dose of study medication and had at least one post-baseline diary assessment.
Measure: Mean (Standard Deviation); unit: SBMs per week
Arm/Group | SP-304 0.3 mg | SP-304 1.0 mg | SP-304 3.0 mg | SP-304 9.0 mg | Placebo
Number analyzed (Participants) | 14 | 14 | 15 | 15 | 20
SBMs per week | 2.4 (2.21) | 4.1 (4.1) | 2.4 (3.39) | 4.2 (2.88) | 2.4 (2.67)

4. Secondary Outcome: Changes From Baseline Overall in Bristol Stool Form Scale (BSFS)
Description: Using a Daily Diary, patients recorded Stool Consistency using the 7-point Bristol Stool Form Scale (BSFS) (1 = separate hard lumps, like nuts; 2 sausage shaped but lumpy; 3 = like a sausage but with cracks on surface; 4 = like a sausage or snake, smooth and soft; 5 = soft blobs with clear-cut edges; 6 = fluffy pieces with ragged edges, a mushy stool; 7 = watery, no solid pieces, entirely liquid). Changes in mean BSFS were assessed from the average 14-day pretreatment baseline to the average during the 2-week treatment period.
Time Frame: Study day 1 through 14
Population: Modified-Intent-to-Treat population: All patients who received at least one dose of study medication and had at least one post-baseline diary assessment. One participant in the SP-304 0.3 mg group did not have post-baseline results.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SP-304 0.3 mg | SP-304 1.0 mg | SP-304 3.0 mg | SP-304 9.0 mg | Placebo
Number analyzed (Participants) | 13 | 14 | 15 | 15 | 20
units on a scale | 1.1 (1.23) | 1.8 (1.18) | 1.6 (1.53) | 1.8 (1.56) | 0.9 (1.23)

5. Secondary Outcome: Changes From Baseline Overall in Ease of Passage (Straining)
Description: Using a Daily Diary, patients recorded Ease of Passage (Straining) using the 7-point Ease-of-Passage Scale (1 = manual disimpaction/enema needed, 2 = severe straining, 3 = moderate straining, 4 = mild straining, 5 = no straining, 6 = urgency, 7 = incontinent). Changes in overall ease of passage (Straining) were assessed from the average 14-day pretreatment baseline to average during the 2-week treatment period
Time Frame: Study Days 1 through 14
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SP-304 0.3 mg | SP-304 1.0 mg | SP-304 3.0 mg | SP-304 9.0 mg | Placebo
Number analyzed (Participants) | 13 | 14 | 15 | 15 | 20
units on a scale | 0.9 (1.05) | 1.6 (1.04) | 1.3 (1.17) | 1.2 (1.06) | 0.5 (1.12)

ADVERSE EVENTS:
Time Frame: 21 Days
Description: Baseline through 14 consecutive days of treatment plus 7 post-treatment days
Arm/Group | SP-304 0.3 mg | SP-304 1.0 mg | SP-304 3.0 mg | SP-304 9.0 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/15 | 0/15 | 1/20
Other Adverse Events (participants affected / at risk) | 3/14 | 6/14 | 2/15 | 6/15 | 4/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SP-304 0.3 mg (N=14) | SP-304 1.0 mg (N=14) | SP-304 3.0 mg (N=15) | SP-304 9.0 mg (N=15) | Placebo (N=20)
Pyelonephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SP-304 0.3 mg (N=14) | SP-304 1.0 mg (N=14) | SP-304 3.0 mg (N=15) | SP-304 9.0 mg (N=15) | Placebo (N=20)
Headache (Nervous system disorders) | 1 | 0 | 0 | 2 | 0
Hyperglycemia (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Bloating (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Hiatus Hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Tingling Feeling in Mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Upset Stomach (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Tiredness (General disorders) | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Elevated Amylase (Investigations) | 1 | 0 | 0 | 0 | 0
Elevated Lipase (Investigations) | 0 | 2 | 1 | 1 | 0
Weight Loss (Investigations) | 0 | 0 | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Intermittent Right Hand Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
One Episode of Neck Muscle Spasm Left Side (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Head Pressure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Intermittent Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dizziness (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Abdominal Cramping (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Excessive Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1
Rhinitis (Due To Pollen) (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Low Back Strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
This Phase 2a study was not sized to evaluate efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the results, either in part or in total (e.g., articles in journals or newspapers, oral presentations, abstracts) by the Investigator(s) or their representative(s), shall require prior notification, review, within a reasonable time frame, and written approval by the Sponsor. Additionally such publications cannot be made in violation of the Sponsor's confidentiality restrictions or to the detriment of the Sponsor's intellectual property rights.